CLINICAL TRIAL: NCT02583906
Title: Sleep Disordered Breathing in Precapillary Pulmonary Hypertension: Effect of CPAP Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S55742
Record Dates: First submitted 2014-04-28; First posted 2015-10-22 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2020-11

CONDITIONS: Sleep-Disordered Breathing; Pulmonary Arterial Hypertension; Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: conditions — Sleep Apnea Syndromes; Pulmonary Arterial Hypertension | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cpap treatment (Other): patients randomized to the 'no cpap' arm will not be treated by CPAP
  Interventions: Device: CPAP
- no cpap (No Intervention): patients randomized to the 'cpap' arm will be treated by CPAP

INTERVENTIONS:
Device: CPAP — Treatment with CPAP for six months in the CPAP arm.
  Other Names: CONTINUOUS POSITIVE AIRWAY PRESSURE
  Arms: cpap treatment

SUMMARY:
Evaluation of the effect of CPAP (continuous positive airway pressure ) treatment in PAH (pulmonary arterial hypertension) and CTEPH (chronic thromboembolic pulmonary hypertension) patients suffering from sleep disordered breathing.

DETAILED DESCRIPTION:
The primary endpoint of the study is to evaluate the effect of CPAP therapy on pulmonary vascular resistance in PAH and CTEPH patients suffering from sleep disordered breathing.

The secondary endpoints are the effect of CPAP on right atrium and right ventricle diameter and ejection fraction measured by echocardiography, 6 minutes walk distance, NYHA class, QOL, endothelial function, sympathetic activity and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years old
* diagnosed with PAH or non-operable CTEPH or operated CTEPH with peristent pulmonary hypertension
* diagnosis of PAH based on cardiac catherisation
* diagnosis of CTEPH confirmed by contrast-enhanced spiral chest CT, pulmonary angiography and V/Q scintigraphy
* recent diagnosis of sleep disordered breathing (polysomnography realized within 3 months before inclusion showing AHI above 15) stable clinical condition for at least 3 months before inclusion as defined by NYHA and a walking distance difference within 10% of the previous 3 months and no change in medical therapy during this 3 months

Exclusion Criteria:

* congenital heart disease
* moderate and severe restrictive or obstructive pulmonary disease with a TLC and a FEV1<60% of the predicted value
* BMI 35kg/m2 or more
* patients already treated with CPAP
* patients with severe sleepiness (epworth sleepiness scale from 18 to 24/24)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-04; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change in PVR (pulmonary vascular resistance) | change in PVR from inclusion at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Catharina Belge, MDPhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium